CLINICAL TRIAL: NCT06318039
Title: Operation ACL: Rehabilitation After Anterior Cruciate Ligament Reconstruction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linnaeus University (Other)
Responsible Party: Principal Investigator, Jesper Augustsson, PhD, Associate Professor, Linnaeus University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB2022-06554-01
Record Dates: First submitted 2024-01-03; First posted 2024-03-19 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novel program (Experimental): Rehabilitation using a novel program
  Interventions: Other: Novel program; Other: Traditional program
- Traditional program (Active Comparator): Rehabilitation using a traditional program
  Interventions: Other: Novel program; Other: Traditional program

INTERVENTIONS:
Other: Novel program — Applying new training method; the Nordic hamstring exercise
Other: Traditional program — Conventional rehabilitation training administered

SUMMARY:
Scientific Research Question

Overall Purpose:

Regarding rehabilitation after anterior cruciate ligament reconstruction (ACLR), there is a knowledge gap - a lack of evidence. Important questions such as how rehabilitation should be structured, what it should include, and how it should be evaluated are currently not clear. Therefore, the investigators plan to conduct a two-year follow-up randomized controlled trial (RCT) on post-ACLR rehabilitation.

Moreover, detailed information on how/under what circumstances the ACL injury occurred is not satisfactorily described in the literature. Therefore, the investigators are planning a new survey that can identify, explain, and prevent the risk factors causing a person to suffer from an anterior cruciate ligament injury.

Specific Objectives:

How should guidelines for rehabilitation after ACLR be structured, what should they include, and how should they be evaluated to best restore knee function in the patient? Can a detailed and comprehensive survey identify, explain, and prevent the risk factors causing a person to suffer from an ACL injury?

DETAILED DESCRIPTION:
The overall aim of the project is to improve the physiotherapeutic guidelines to enhance the quality of rehabilitation for patients with surgically repaired anterior cruciate ligament (ACL) injuries. ACL injury is a severe knee injury that often prevents young individuals from continuing sports activities at their desired level. It can eventually lead to knee osteoarthritis within 10-15 years after the initial injury. Despite existing research on preventive training for young athletes in high-risk sports such as soccer, handball, and floorball, this injury remains common. ACL injury in young female athletes engaged in contact sports is 2-5 times more prevalent compared to young males. Regarding rehabilitation after ACL reconstruction, literature often indicates inadequacies where full muscle strength or jumping ability has not been regained. Despite this, patients often return to sports activities, which may increase the risk of re-injury. Guidelines for structuring rehabilitation, its content, and evaluation need improvement accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Athletes or recreational athletes that have undergone ACLR

Exclusion Criteria:

* Patients that have undergone ACLR that are nor athletes or recreational athletes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Isokinetic muscle strength | Tests at 8, 12, 18 and 24 months post-ACLR.
  Test of each patient's unilateral maximal isokinetic muscle strength for the involved and the uninvolved leg, using an isokinetic dynamometer (Biodex isokinetic dynamometry system 4).
Single-leg hop performance | Tests at 8, 12, 18 and 24 months post-ACLR.
  Test of each patient's single-leg hop performance for the involved and the uninvolved leg. The goal is to have a less than 10% difference in hop distance between the injured limb and uninjured limb.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Survey at 10 weeks and 8, 12, 18 and 24 months post-ACLR.
  Knee Injury and Osteoarthritis Outcome Score (KOOS) evaluates both short-term and long-term consequences of knee injury. It holds 42 items in 5 separately scored subscales; Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL). The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.
ACL Return to Sport after Injury scale | Survey at 10 weeks and 8, 12, 18 and 24 months post-ACLR.
  The ACL - Return to Sport after Injury (ACL-RSI) scale measure athletes' emotion, confidence, and risk appraisal when returning to sports after an ACL injury and/or reconstructive surgery. The survey consists of 12 items that are graded on a visual analogue scale from 0 points (extremely negative psychological responses) to 100 points (no negative psychological responses).

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Augustsson, PhD, Principal Investigator — Linneuniversitetet
Locations (1):
- Linnaeus University, Kalmar, Sverige, Sweden

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make individual participant data (IPD) available to other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From year 2026 to 2031.
Access Criteria: Other researcher within the field of ACLR-rehabilitation.

REFERENCES:
- See also: The project's homepage — https://lnu.se/en/research/research-projects/project-operation-acl/